CLINICAL TRIAL: NCT00599313
Title: Phase II Trial of Sunitinib Malate for the Therapy of Progressive Metastatic Androgen Independent Prostate Cancer (AIPC) Following Docetaxel-based Chemotherapy
Brief Title: Phase II Sunitinib Prog Met AIPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05112; 2006-0012 (Other: Pfizer)
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate (Experimental): Sunitinib Malate (Sutent) (50 mg/day on Days 1-28 of 42-day cycles)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50 mg/day orally each of Days 1-28 of each 6 week cycle
  Other Names: Sunitinib malate; Sutent

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) Sutent has on you and your prostate cancer.

DETAILED DESCRIPTION:
The following rationale can be made for a Phase II trial to evaluate sunitinib malate (Sutent) for the therapy of progressive metastatic androgen-independent prostate cancer (AIPC) following prior docetaxel chemotherapy. Since most patients with metastatic AIPC following prior chemotherapy clinically progress rapidly, we believe that achieving a 30% freedom from clinical progression (PFS) (not including PSA progression) at 12 weeks represents biologically active therapy. Sunitinib malate (Sutent) represents a tolerable and convenient form of therapy with the potential for improving outcomes in AIPC.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this study if he meets all of the following criteria:
* Histologically confirmed, adenocarcinoma of the prostate
* Stage IV(metastatic) disease, documented on CT, MRI, or X-ray
* Progressive disease (PSA or clinical): PSA progression defined as baseline increase followed by any serial increase after 2 weeks; clinical progression by symptomatic or radiologic criteria.
* An elevated PSA level of for patients progressing by PSA criteria is required
* Currently on androgen ablation hormone therapy (an LHRH agonist or orchiectomy) with testosterone level <50ng/dL)
* Has received 1 or 2 prior chemotherapy regimens (no more than 2). One prior regimen must be docetaxel.
* Has an ECOG Performance Status (PS) 0-2
* Is greater than 18 years of age
* Meets protocol defined laboratory values
* Has adequate cardiac function in the opinion of the Investigator
* Has no uncontrolled arrhythmia or hypertension
* Resolution of all acute toxic effects of prior chemotherapy or surgical procedures to NCI CTCAE Version 3.0 Grade less than 1, in the opinion of the Treating Physician
* If fertile, patient has agreed to use an acceptable method of birth control to prevent pregnancy for the duration of the study and for a period of 2 months thereafter
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

* A patient will be excluded from this study if he meets any of the following criteria:
* Has any disease other than that described in inclusion criterion #1
* Had prior treatment with Sutent
* Has not received prior docetaxel for the current disease
* Has received any prior radionuclide therapy
* Has received prior radiation to >50% of the bone marrow
* Is receiving concurrent immunotherapy
* Has a history of hypersensitivity to any of the components of Sutent: mannitol, croscarmellose sodium, povidone (K-25) and magnesium stearate as inactive ingredients. The orange gelatin capsule shells contain titanium dioxide, and red iron oxide. The caramel gelatin capsule shells also contain yellow iron oxide and black iron oxide. The printing ink contains shellac, propylene glycol, sodium hydroxide, povidone and titanium dioxide.
* Has had significant bleeding in previous 4 weeks
* Has had any of the following within the prior 6 months: severe/unstable angina, myocardial infarction, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident, transient ischemic attack, or pulmonary embolism
* Is receiving concurrent bisphosphonate therapy; long-standing bisphosphonate therapy (initiated >8 weeks prior to registration) is acceptable. Bisphosphonates started within the prior 8 weeks will not be allowed since this may affect other study endpoints and render their interpretation difficult
* Has received treatment with radiation therapy, surgery, chemotherapy, ketoconazole, corticosteroids, or an investigational agent within 4 weeks prior to registration, (6 weeks for radiation therapy, nitrosureas or Mitomycin C)
* Has uncontrolled arrhythmia or hypertension
* Has evidence of uncontrolled CNS involvement (previous radiation and off steroids is acceptable)
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin), which could affect the diagnosis or assessment of any of the study drugs
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — US Oncology Research
Locations (45):
- United States (45):
  - Hematology Oncology Associates, Phoenix, Arizona
  - Connecticut Oncology & Hematology, LLP, Torrington, Connecticut
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Care & Hematology Specialista of Chicagoland, Niles, Illinois
  - Hope Center, Terre Haute, Indiana
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Alliance Hematology Oncology PA, Westminster, Maryland
  - Missouri Cancer Associates, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Arch Medical Services, Inc. DBA The Cntr for Cancer Care & Research, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NH Oncology-Hematology PA, Hooksett, New Hampshire
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Interlakes Oncology Hematology, PC, Rochester, New York
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Cancer Center-Abilene(South), Abilene, Texas
  - Texas Oncology, P.A.-Amarillo, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, P.A.-Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Onclogy, P.A., Dallas, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology-Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - HOAST-Medical Dr., San Antonio, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Texas Oncology Cancer Care and Research, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 36
Completed | 0
Not Completed | 36
Not completed — Adverse Event | 19
Not completed — Disease Progression | 12
Not completed — Patient Request | 4
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: Total participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 32
  Black | 3
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS) Time at 1-year.
Description: PFS is measured from the date of registration to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 12 months
Population: ITT population
Measure: Median (Full Range); unit: weeks
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 36
weeks | 19.4 [2.6 to 48.3]

2. Secondary Outcome: Overal Survival (OS) Rate at 1-year.
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 12 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Probability of Survival at 1-year
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 36
Probability of Survival at 1-year | 0.42 [0.23 to 0.60]

3. Secondary Outcome: Prostate Specific Antigen (PSA) Response
Description: Percentage of participants whose PSA value declined to 50% when compared to the value at the baseline.
Time Frame: Baseline and up to 12 months
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 33
percentage of participants | 12.1 [3.4 to 28.2]

4. Secondary Outcome: Change of PSA Doubling Time
Description: Difference of PSA doubling time between baseline and end of the treatment.
Time Frame: Baseline and up to 12 months
Population: Patients who had measurements of prior and post doubling time.
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 25
months | 0.5 [-5.1 to 43.7]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR = Complete Response (CR) + Partial response (PR). CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: 12 months
Population: Only patients with baseline measurable lesions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 18
percentage of participants | 11.1 [1.4 to 34.7]

6. Secondary Outcome: Percentage of Participants With Decrease in Present Pain Intensity (PPI) From Baseline.
Description: Pain score decreased >=2 points from baseline. The PPI scale has the following descriptors: 0=no pain, 1=mild pain, 2=discomforting pain, 3=distressing pain, 4=horrible pain, and 5=excruciating pain. The patient will be asked to self-assess and record their PPI in the study diary. Upon diary review, the study nurse will utilize the PPI daily scores to calculate the week's average. The weekly PPI score during the study is the average of the daily PPI scores, based on a minimum of 3 daily PPI assessments during a week's period.
Time Frame: Baseline and up to 12 months
Population: Patients with pain measurement at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 22
percentage of participants | 13.6 [6.3 to 20.9]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treated patients only, assessed at each treatment visit.
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 7/35
Other Adverse Events (participants affected / at risk) | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=35)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (2)
FAILURE KIDNEY ACUTE (Renal and urinary disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
STROKE (Vascular disorders) | 1 (1)
THROMBOSIS PULMONARY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=35)
ALKALINE PHOSPHASTASE SERUM INCREASE (Metabolism and nutrition disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 13 (17)
ANOREXIA (Gastrointestinal disorders) | 13 (18)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 11 (13)
DYSGUESIA (Gastrointestinal disorders) | 3 (3)
EDEMA (Blood and lymphatic system disorders) | 2 (2)
FATIGUE (General disorders) | 16 (25)
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 3 (3)
HYPERTENSION (Vascular disorders) | 3 (3)
LEUCOPENIA (Blood and lymphatic system disorders) | 5 (14)
MALAISE (General disorders) | 2 (2)
MUCOSITIS (Gastrointestinal disorders) | 6 (9)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 12 (20)
NEUROPATHY (Nervous system disorders) | 2 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 11 (16)
RASH (Skin and subcutaneous tissue disorders) | 6 (6)
STOMATITIS (Gastrointestinal disorders) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (8)
VOMITING (Gastrointestinal disorders) | 5 (5)
WEIGHT LOSS (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No